CLINICAL TRIAL: NCT02798393
Title: Randomized Double-Blind Study of the Efficacy of Near Infrared Phototherapy on Sensation and Pain in Type 2 Diabetic Neuropathy
Brief Title: Efficacy of Near Infrared Phototherapy in Type 2 Diabetic Neuropathy
Acronym: ResearchNIR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study blind compromised.
Sponsor: Healthlight, LLC (Industry)
Collaborators: Clin-Assist, LLC (Unknown); Midwest Medical Research (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIR-001
Record Dates: First submitted 2016-06-04; First posted 2016-06-14 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-02

CONDITIONS: Neuropathy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- HL-Sham (Sham Comparator): The placebo device (also referred to as the HL-SHAM device) will have an identical appearance to the HL-NIR device. Though the HL-NIR device will be applied, there will be no treatment administered.
  Interventions: Other: Sham
- HL-NIR (Experimental): The device referred to as the HL-NIR device includes both a podiatric or foot and leg component, similar to a loose fitting boot, that is easily applied to all subjects (one size fits all). Application of the device is snug but comfortable without risk for constriction of soft tissue.
  Interventions: Other: Infrared Phototherapy

INTERVENTIONS:
Other: Infrared Phototherapy — Subjects will wear a cuff on their extremities for a set period of time at set intervals over a period of several weeks. The cuff will emit the Infrared Phototherapy treatment (or sham if randomized to the non-treat group).
  Arms: HL-NIR
Other: Sham
  Arms: HL-Sham

SUMMARY:
This is a double blind, randomized, placebo-controlled study in which a total of 120 patients will be selected from a broad spectrum group of typical Americans (all demographics including various races and both genders as well as ages from 25-90) who have confirmed Type 2 Diabetes Mellitus and suffer from mild to moderate lower extremity Peripheral Neuropathy. All patients will meet inclusion and/or exclusion criteria.

DETAILED DESCRIPTION:
This is a double blind, randomized, placebo-controlled study in which a total of 120 patients will be selected from a broad spectrum group of typical Americans (all demographics including various races and both genders as well as ages from 25-90) who have confirmed Type 2 Diabetes Mellitus and suffer from mild to moderate lower extremity Peripheral Neuropathy. All patients will meet inclusion and/or exclusion criteria.

Randomization and Application of HL Device The placebo controlled group of 60 patients will be randomized from the group of 120 patients by one designee who selects the placebo vs treatment groups based on acceptable statistical standards for determining placebo vs treatment arms of research studies. There will be two different HL Devices. There will be the HL-NIR device that includes NIR diodes and performs Near Infrared therapy and an identical appearing second device, the HL-SHAM device, that is used as the placebo device and although appearance is identical, this device does not perform Near Infrared treatment. Both placebo group and treatment group subjects will have the NIR or sham device applied to both lower extremities for a short duration three times a week over the course of several weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of Type 2 Diabetes Mellitus on oral hypoglycemic medication, and/or injectable insulin
2. Hg A1C 5.7 or above ((Pre-Diabetes is 5.7 to 6.4%) (Diabetes is above 6.5%)), Hg A1C below 9.1
3. Peripheral Neuropathy of the feet, or feet and legs
4. If the patient has a lower extremity ulceration that is not showing any signs of infection, and this patient has ABPI and TBPI above 55 mm of Hg, they may be included in the study, at the discretion of the Principal Investigator (PI). If the patients infection is localized (not osseous in nature) and the infection can be treated and cleared and remain uninfected for 30 days, the patient could be reevaluated and included in the study at the discretion of the PI.
5. If the patient has an area of injury or erythema or induration, they may still be included in the study if they have ABPI and TBPI above 55 mm of Hg, at the discretion of the PI
6. Positive MNS
7. All medications or other treatments for neuropathy are held constant for at least 30 days prior to the study, during the baseline and treatment period of the study.
8. Subjects will have pain and insensate sites on each foot (both feet will be assessed and pain scales for both extremities will be measured/followed).
9. Moderately positive MNS score.

Exclusion Criteria:

1. Any other causes of Peripheral Neuropathy
2. Known Spinal Stenosis
3. Previous Back Injury
4. Comorbid issues of exacerbated CHF
5. Exacerbation of COPD
6. Chronic steroid use
7. Underlying connective tissue disease
8. Previous trauma or underlying fracture
9. Current injury or trauma
10. Skin ulceration
11. ABPI and TBPI measurements will be measured and if the patient has an open ulceration with signs of infection and the wound is weeping any serous or purulent fluid, anywhere on their foot or lower extremity
12. Negative MNS
13. Previous amputation of a portion of the foot
14. Amputation of digit or digits are not considered exclusion criteria
15. Previous arterial bypass graft
16. Known cardiac arrhythmia
17. HG A1C above 9.1%
18. Uncontrolled fasting blood sugar, or Type 1 Diabetes.
19. If on any anti-epileptic or anti-depressant medications
20. If patient has had any change in pain or anti-inflammatory medication anytime within the past 30 days.
21. Pregnancy or planned pregnancy (If a patient has begun our research study and does not know that they are pregnant or they become pregnant during the study, they will not be dropped from the study) (Reasoning: there is no evidence for or against using HealthLight therapy in pregnant individuals.)
22. Active osteomyelitis or positive for osteomyelitis within the past six months
23. Open ulceration with signs and symptoms of active infection.
24. Known Peripheral Arterial Disease (PAD)
25. Previous Lumbar surgery or Lumbar Disc intervention anytime within the past year

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Decrease in Pain (MPI Pain Scale) | 90 Days
  Decrease in pain as measured by the Multidimensional Pain Inventory (MPI) pain scale

SECONDARY OUTCOMES:
Improvement in Sensation | 90 Days
  Improvement in sensation as measured by Michigan Neuropathy Screening (MPS) scoring

OTHER OUTCOMES:
Safety Assessment (incidence of treatment related AEs at each follow up visit) | 90 Days
  Incidence of treatment related adverse events at each follow up visit

CONTACTS AND LOCATIONS:
Overall Officials: Kipp Van Camp, DO, Principal Investigator — Midwest Medical Research
Locations (1):
- Midwest Medical Research, Topeka, Kansas, United States

IPD SHARING:
Plan to Share IPD: No